CLINICAL TRIAL: NCT03360656
Title: Transnasal Induction of Normothermia in Febrile Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CoolTech LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00074620
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Fever; Seizures; Metabolic Encephalopathy
Keywords: shivering, fever, normothermia
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Fever; Seizures; Brain Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transnasal Thermal Regulating Device (Experimental): Consented subjects will undergo cooling via transnasal thermal regulating device for a period of 8 to 24 hours
  Interventions: Device: Transnasal Thermal Regulating Device

INTERVENTIONS:
Device: Transnasal Thermal Regulating Device — Placement of transnasal thermal regulating device to reduce temperature in febrile patients for a period of 8 to 24 hours

SUMMARY:
The objective of this study is to evaluate safety and performance of the COOLSTAT® Transnasal Thermal Regulating Device in reducing temperature in a population of febrile subjects who meet the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the Neurosciences Critical Care Unit (NCCU).
2. Patient has ischemic or hemorrhagic stroke, seizure, or metabolic encephalopathy.
3. Patient is orally intubated or has tracheostomy tube and is mechanically ventilated.
4. Planned stay in NCCU > 24 hours.
5. Must have informed consent from the patient or the legally authorized representative (LAR)

Exclusion Criteria:

1. Age < 18 years old or > 95 years.
2. Intubation is contraindicated.
3. With a coagulopathy. INR above 1.5 or PTT above 45 seconds.
4. Hemodynamic instability, including elevated SPB for >5 minutes despite standard of care interventions (SPB ≥ 160 mmHg for intracerebral hemorrhagic stroke; SPB ≥ 220 mmHg for subarachnoid hemorrhagic stroke or ischemic stroke).
5. History of cryoglobulinemia.
6. History of sickle cell disease.
7. History of serum cold agglutinin disease.
8. Active/ongoing of nose bleeds.
9. Known or suspected pregnancy.
10. Participation in another ongoing investigational study.
11. Prisoners and/or patients for whom no LAR is available.
12. Patient is in airborne/droplet disease isolation protocol.
13. Patient is or suspected to be immunocompromised;
14. Low platelet count defined as < 100k (thrombocytopenia).
15. Nasal septal deviations (per CT scan; any degree).
16. Chronic rhinosinusitis.
17. Prior skull-based surgery
18. Penetrating cranial trauma.
19. Recent nasal trauma or anterior base skull fracture.
20. Presence of cardiac arrhythmias including: sustained tachycardia defined as heart rate above 120 beats per minute, or sustained bradycardia defined as heart rate below 60 beats per minute.
21. Refractory hypoxemia defined as partial pressure of oxygen in arterial blood (paO2) below 60 torr or oxyhemoglobin saturation below 90% despite endotracheal intubation, mechanical ventilation, and provision of supplemental oxygen of up to 0.60.
22. Refractory hypercarbia defined as partial pressure of carbon dioxide in arterial blood (paCO2) above 50 torr despite endotracheal intubation and conventional mechanical ventilation.
23. History of cardiac arrhythmia as listed above.
24. BMI of ≤ 15 kg/m2 or ≥ 40kg/m2

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Badjatia, MD MS, Principal Investigator — Univ of Maryland
Locations (3):
- United States (3):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Texas, Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnold S, Armahizer M, Torres LF, Tripathi H, Tandri H, Chang JJ, Choi HA, Badjatia N. Minimizing Shivering During Targeted Normothermia: Comparison Between Novel Transnasal and Surface Temperature-Modulating Devices. Neurocrit Care. 2023 Dec;39(3):639-645. doi: 10.1007/s12028-023-01793-3. Epub 2023 Jul 27. PMID 37498457

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transnasal Thermal Regulating Device
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 30
Arm/Group | Transnasal Thermal Regulating Device
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.93 (15.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 9
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Cooling Performance
Description: Ability of transnasal thermal regulating device to reduce core body temperature within 4 hours of initiation
Time Frame: 4 hours
Population: The primary efficacy analysis for cooling performance will be based on the evaluable populations of subjects who undergo cooling treatment with the COOLSTAT System. Analysis will be performed on treatment initiated and treatment completed populations. Subjects who achieve normothermia (core temperature ≤ 37.5 °C) within 4 hours of starting COOLSTAT treatment and maintain normothermia for the duration of the treatment will be determined to have been treated successfully.
Measure: Count of Participants; unit: Participants
Arm/Group | Transnasal Thermal Regulating Device
Number analyzed (Participants) | 30
Participants | 19

ADVERSE EVENTS:
Time Frame: Adverse events were collected during a 48 hour period, starting when the subject was placed on CoolStat, during the 24 hour cooling period, and for the 24 hour post-cooling observation period.
Arm/Group | Transnasal Thermal Regulating Device
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 15/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transnasal Thermal Regulating Device (N=30)
Shivering (Nervous system disorders) | 9 (11)
Insufficient cooling (Nervous system disorders) | 5 (5)
Adverse effects on systemic blood pressure (Cardiac disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT03360656/Prot_SAP_000.pdf